CLINICAL TRIAL: NCT02374632
Title: Gut Hormones as Mediators of Different Weight Loss Responses After Roux-en-Y Gastric Bypass
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Kirstine Nyvold Bojsen-Moeller, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KBM-R2-14
Record Dates: First submitted 2015-02-17; First posted 2015-03-02 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Bariatric Surgery (Gastric Bypass); Severe Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low EBL (Other): Gastric bypass operated patients with low postoperative excess body weight loss (EBL) <50%.
  Interventions: Meal tests after saline/octreotide injection in a randomized order, sham feeding.
  Interventions: Other: Meal tests after saline injection; Other: Meal tests after octreotide injection; Other: Sham feeding
- High EBL (Other): Gastric bypass operated patients with high postoperative excess body weight loss (EBL) >70% matched with respect to age, gender and preoperative BMI in the LowEBL group.
  Interventions: Meal tests after saline/octreotide injection in a randomized order, sham feeding.
  Interventions: Other: Meal tests after saline injection; Other: Meal tests after octreotide injection; Other: Sham feeding

INTERVENTIONS:
Other: Meal tests after saline injection — Fixed breakfast meal and ad libitum lunch meal
Other: Meal tests after octreotide injection — Fixed breakfast meal and ad libitum lunch meal
Other: Sham feeding

SUMMARY:
After gastric bypass, 10-20% of patients will obtain a suboptimal weight loss, often defined as <50% of the excess body weight. Exaggerated meal related secretion of gut hormones seem important for appetite reduction and subsequent weight loss after gastric bypass, however it is not clear whether different gut hormone responses are responsible for different postoperative weight loss responses. The purpose of the study is to investigate gut hormone secretion, vagal integrity and the effect of octreotide on ad libitum food intake in patients with suboptimal weight loss after gastric bypass and compare results to a matched group of gastric bypass operated patients with high postoperative weight loss but similar age, sex and preoperative BMI.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated primary Roux-en-Y gastric bypass >12 months ago
* Postoperative weight loss of >60%EBL or <50%EBL.

Exclusion Criteria:

* Inadequately treated thyroid disease
* Hemoglobin <6.5 mM
* Pregnancy or breastfeeding

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Glucagon-like peptide-1 (GLP-1) secretion (Between groups difference in incremental Area-under-the curve (iAUC) GLP-1 after fixed breakfast meal on saline day) | 0-240 min
  Between groups difference in iAUC GLP-1 after fixed breakfast meal on saline day
Peptide YY (PYY) secretion (Between groups difference in iAUC PYY after fixed breakfast meal on saline day) | 0-240 min
  Between groups difference in iAUC PYY after fixed breakfast meal on saline day
Ghrelin secretion (Between groups difference in iAUC Ghrelin after fixed breakfast meal on saline day) | 0-240 min
  Between groups difference in iAUC Ghrelin after fixed breakfast meal on saline day

SECONDARY OUTCOMES:
Ad libitum food intake | 240 min
  Between groups difference in ad lib food intake
Effect of octreotide on Ad libitum food intake (Between groups difference in %change in ad lib food intake between saline and octreotide day) | 240 min
  Between groups difference in %change in ad lib food intake between saline and octreotide day
Vagal insufficiency (Between groups difference in % change in pancreatic polypeptide (PP) from fasting to early peak levels (15-30 min) after sham feeding) | 0-30 min
  Between groups difference in % change in PP from fasting to early peak levels (15-30 min) after sham feeding

OTHER OUTCOMES:
Appetite scores (Between groups differences in VAS scores after meal test and sham feeding test) | 0-240 min, 240-270 min, 0-75 min
  Between groups differences in VAS scores after meal test and sham feeding test
Genetic profile (Between groups differences in gene variants investigated with a HumanCoreExome chip) | 0 min
  Between groups differences in gene variants investigated with a HumanCoreExome chip
Gut microbiota (Between groups differences in gut microbiome investigated with next generation sequencing) | feces sample at home before intervention
  Between groups differences in gut microbiome investigated with next generation sequencing
Food intake (Between groups differences in food intake evaluated by questionnaires and diet registration) | 4 weeks questionnaires and 4 days of registration
  Between groups differences in food intake evaluated by questionnaires and diet registration
Physical activity (Between groups differences in food intake evaluated by questionnaires and accelerometer) | 4 weeks questionnaires and14 days of registration
  Between groups differences in food intake evaluated by questionnaires and accelerometer

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Hvidovre Hospital, Hvidovre, Denmark